CLINICAL TRIAL: NCT01714063
Title: Drug Delivery Via Pressurized Metered-dose Inhaler and Valved Holding Chamber in Asthmatic Children: Determination of Delivered Dose Following Coordinated and Uncoordinated Use
Status: Completed | Type: Observational
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: RDD-2010-001
Record Dates: First submitted 2012-10-18; First posted 2012-10-25 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: pediatric; asthma; metered dose inhaler; valved holding chamber; pMDI; VHC
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Age 5-6.5: Group 1 will consist of 16 children aged 5-6.5 years
  Interventions: Device: Pressurized Metered-Dose Inhaler
- Aged 6.6- 8 years: Group 2 will consist of 16 children aged 6.6- 8 years
  Interventions: Device: Pressurized Metered-Dose Inhaler

INTERVENTIONS:
Device: Pressurized Metered-Dose Inhaler — Pressurized Metered-Dose Inhaler

SUMMARY:
The primary objective of this study is to determine ex vivo the amount of fluticasone deposited onto a filter (delivered dose) interposed between the OptiChamber Diamond Valved Holding Chamber (VHC) mouthpiece and the subject's mouth during coordinated and uncoordinated actuation/inhalation maneuver.

ELIGIBILITY:
Inclusion Criteria:

* • Asthmatic children between the ages of 5 and 8 followed at Arkansas Children's Hospital.

  * The subjects must be available to complete the study.
  * The subject's parent(s) and/or the subject's legal guardian must provide written informed consent to participate in the study.
  * The subject must provide assent when older than 7 years old.
  * The subjects should have used a pMDI VHC previously and be able to use a VHC with mouthpiece.
  * The subjects should have been prescribed fluticasone or another inhaled corticosteroid delivered via a pMDI VHC combination.
  * Clinically stable asthma.
  * Cooperative, i.e., subject should be able to follow and understand instructions.
  * The subject must satisfy the study investigator about his/her fitness to participate in the study.

Exclusion Criteria:

* Clinically significant respiratory disease in the previous 4 weeks.
* Participation in any other clinical trial in the previous 4 weeks.
* Lack of cooperation, subject cannot follow and understand instructions.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 40 subjects aged 5-8 diagnosed with asthma
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Berlinski, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Berlinski A, von Hollen D, Pritchard JN, Hatley RH. Delay Between Shaking and Actuation of a Hydrofluoroalkane Fluticasone Pressurized Metered-Dose Inhaler. Respir Care. 2018 Mar;63(3):289-293. doi: 10.4187/respcare.05782. Epub 2017 Nov 21. PMID 29162718
- [Derived] Berlinski A, von Hollen D, Hatley RHM, Hardaker LEA, Nikander K. Drug Delivery in Asthmatic Children Following Coordinated and Uncoordinated Inhalation Maneuvers: A Randomized Crossover Trial. J Aerosol Med Pulm Drug Deliv. 2017 Jun;30(3):182-189. doi: 10.1089/jamp.2016.1337. Epub 2016 Dec 15. PMID 27977309

RESULTS

PARTICIPANT FLOW:
Groups:
- Pressurized Metered-Dose Inhaler: All participants that were consented to use the Pressurized Metered-Dose Inhaler in this study were considered.
Period: Overall Study
Arm/Group | Pressurized Metered-Dose Inhaler
Started | 34
Completed | 32
Not Completed | 2
Not completed — Equipment malfunction | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants that were consented to the study were considered.
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.4 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 15
Height [Mean (Standard Deviation); unit: centimeters] | 119.3 (7.7)
Weight [Mean (Standard Deviation); unit: kilograms] | 26.4 (8.6)
Time Using Valved Holding Chamber [Mean (Standard Deviation); unit: years] | 3 (2.5)
Previous Mouthpiece Experience [Mean (Standard Deviation); unit: percentage of participants] | 13 (41)

OUTCOME MEASURES:

1. Primary Outcome: Delivered Dose of Fluticasone (on the Filter)
Description: This is a measure of the the amount of fluticasone deposited onto a filter (delivered dose) during coordinated and uncoordinated actuation/inhalation maneuver. The coordinated maneuver occurs when the firing of the fluticasone is coordinated with the inhalation of the patient . An uncoordinated maneuver occurs when the firing of the fluticasone is coordinated with the exhalation of the patient.
Time Frame: Day 1
Measure: Mean (99% Confidence Interval); unit: Percent filter dose of fluticasone
Arm/Group | Age 5-6.5 | Aged 6.6- 8 Years
Number analyzed (Participants) | 16 | 16
Percent filter dose of fluticasone
  Coordinated | 48 [44 to 52] | 45 [39 to 51]
  Uncoordinated | 41 [36 to 47] | 40 [35 to 45]
Statistical Analysis 1: Comparison: Age 5-6.5 vs Aged 6.6- 8 Years; Test type: Other — We used a paired T-test for statistical analysis to compare the filter dose. Using the 1% significance level and assuming a between-subject standard deviation of 60 lg (27%) for the difference between coordinated and doses, 32 subjects are sufficient to detect a 45 lg (20%) difference with 95% confidence.uncoordinated filter; p < 0.001, paired t-test

2. Primary Outcome: Delivered Dose of Fluticasone (on the Filter) Comparing Coordinated and Uncoordinated Maneuvers
Description: as for outcome 1
Time Frame: Day 1
Population: 1 participant was excluded from the filter data because they were an outlier
Measure: Mean (99% Confidence Interval); unit: Percent filter dose of fluticasone
Groups:
- All Participants: Data among all participants were compared for the coordinated and uncoordinated effort
Arm/Group | All Participants
Number analyzed (Participants) | 31
Percent filter dose of fluticasone
  Coordinated | 46 [43 to 50]
  Uncoordinated | 41 [37 to 44]

3. Secondary Outcome: Inspiratory Peak Flow
Description: Inspiratory peak flow is a person's maximum speed of inspiration, as measured with a peak flow meter, a small, hand-held device used to monitor a person's ability to breathe in air.
  This study compared the inspiratory peak flows of all participants between the coordinated and uncoordinated maneuvers.
Time Frame: Day 1
Population: 1. participant was excluded from both the coordinated because of their breathing profile
  2. participants were excluded from the uncoordinated effort because of their breathing profile
Measure: Mean (99% Confidence Interval); unit: L/min
Groups:
- Coordinated Effort: Data among all participants were compared for the coordinated maneuver.
- Uncoordinated Effort: Data among all participants were compared for the uncoordinated maneuver.
Arm/Group | Coordinated Effort | Uncoordinated Effort
Number analyzed (Participants) | 31 | 30
L/min
  1st Breath | 25.2 [20.5 to 30] | 22.8 [17.6 to 28.1]
  2nd Breath | 23.3 [18.5 to 28.1] | 22 [17.3 to 26.6]
  3rd Breath | 23.2 [18.3 to 28] | 22.5 [17.1 to 27.9]
  All Breaths | 23.9 [21.3 to 26.5] | 22.4 [19.6 to 25.2]

4. Secondary Outcome: Inspiratory Tidal Volume
Description: Inspiratory tidal volume is a person's lung volume representing the normal volume of air displaced between normal inhalation and exhalation when extra effort is not applied. In a healthy, young human adult, tidal volume is approximately 500 mL per inspiration or 7 mL/kg of body mass.
  This study compared the inspiratory tidal volume of all participants between the coordinated and uncoordinated maneuvers.
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (99% Confidence Interval); unit: mL
Arm/Group | Coordinated Effort | Uncoordinated Effort
Number analyzed (Participants) | 31 | 30
mL
  1st Breath | 286 [209 to 363] | 269 [212 to 362]
  2nd Breath | 281 [215 to 363] | 259 [186 to 333]
  3rd Breath | 302 [227 to 378] | 266 [201 to 331]
  All | 291 [250 to 332] | 271 [228 to 314]

5. Other Pre Specified Outcome: Measurement Residual Amount of Drug (Fluticasone) Deposited Within the OptiChamber Diamond VHC
Description: Collect the residual amount of drug (fluticasone) deposited within the OptiChamber Diamond VHC by washing the internal surfaces of the VHC and the Pressurized Metered Dose Inhaler (pMDI) boot
Time Frame: Day 1
Population: This is a measure of an inhaler study, not a nebulizer study. Therefore this data was not collected or analyzed as it would not be applicable to this type of study.
Arm/Group | Coordinated Effort | Uncoordinated Effort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No